CLINICAL TRIAL: NCT05186948
Title: Development and Validation of a Novel Functional Eye-Tracking Software Application for Cancer-related Cognitive Impairment (CRCI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Innodem Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ETNA-CRCI
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cancer-related Cognitive Impairment
Keywords: Cancer-related cognitive impairment (CRCI); Eye Movement Biomarkers; Eye-tracking
MeSH Terms: interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients (stages I-IIIA): 200 patients with an initial diagnosis of breast cancer stages I-IIIA and scheduled chemotherapy, fulfilling the eligibility criteria
  Interventions: Device: Eye-Tracking
- healthy control: Group of 30 healthy control participants, matched for age and sex, with no evidence or history of significant neurodegenerative disorder affecting brain function.
  Interventions: Device: Eye-Tracking

INTERVENTIONS:
Device: Eye-Tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
This study aims to develop and validate a sensitive and non-invasive eye-tracking software application.

DETAILED DESCRIPTION:
This study will obtain participant responses to brief cognitive tests designed to evaluate several key functions known to be affected by the Cancer-related cognitive impairment (CRCI) and non-invasive eye movement measurements in response to visually presented stimuli during specifically designed eye-tracking tests. The study data will be used to develop machine learning algorithms and validate a software application intended to track the progressive component of the Cancer-related cognitive impairment (CRCI) and associated cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  1. Able to provide informed consent.
  2. Visual acuity sufficient to be able to read the consent form with corrective lenses.
  3. Over 18 years of age.
  4. English- or French-speaking.
* For patients only:

  1. Initial diagnosis of breast cancer stage I-IIIA and scheduled chemotherapy
  2. First-time cancer diagnosis.
  3. ECOG performance < 2
  4. Receiving curative intent chemotherapy: either Adriamycin/Cyclophosphamide for 4 cycles followed by weekly Taxol for 12 cycles or Taxotere/Cyclophosphamide for 4 cycles

Exclusion Criteria:

* For all participants:

  1. Evidence or medical history of neurological/psychiatric issues known to affect movements and oculomotor control.
  2. Presence of comorbid neurological conditions to avoid eye movement anomaly confounds (Strabismus, cranial nerve palsy, stroke-causing hemianopsia).
  3. Diagnosis of macular edema or other pre-existing ocular conditions that would prevent participants from performing the eye movement assessments.
  4. Previous history of cancer or chemotherapy
  5. Distant metastases
  6. Recent (less than three months from enrollment) start of, change of dose, or irregular use of, new prescription drugs known to influence ocular motor visual function, such as benzodiazepines, antipsychotics and anticonvulsants. Occasional use of benzodiazepines for medical procedures is permitted, at the investigator's discretion, but should not occur within a short time period prior to or during an eye movement assessment.
  7. Diagnosis of a substance abuse disorder.
  8. Recreational drug use (e.g., alcohol, marijuana) is a potential exclusion criterion that will be determined on an individual basis as per the discretion of the research team. All recreational drug use will be documented.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be obtained from 200 patients with an initial diagnosis of breast cancer stages I-IIIA and scheduled chemotherapy, fulfilling the eligibility criteria. Data will also be acquired from a group of 30 healthy control participants. Groups will be matched for age and sex.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Symbol Digit Modalities Test (SDMT) score at Month 36 | Baseline and Month 36
  The SDMT is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Scoring involves summing the number of correct substitutions within the 90 second interval.

SECONDARY OUTCOMES:
Change from Baseline in The Controlled Oral Word Association Test (COWAT) scores at Month 36 | Baseline and Month 36
  The Controlled Oral Word Association Test from the Halstead-Reitan Neuropsychological Battery is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds).
Change from Baseline in The Trail Making Test (TMT) Parts A & B scores at Month 36 | Baseline and Month 36
  The Trail Making Test (TMT) is a neuropsychological test that provides information on visual search, scanning, speed of processing, mental flexibility and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
Change from Baseline in The Hopkins Verbal Learning Test-Revised (HVLT-R) scores at Month 36 | Baseline and Month 36
  The Hopkins Verbal Learning Test (HVLT-R) is a neuropsychological test that provides information on verbal learning and memory. The assessment consists of memorization of a list of words to test the ability to recall immediately after memorization (immediate recall) and after a 20-minute delay (delayed recall).

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center-Cedar Cancer Center, Montreal, Quebec, Canada